CLINICAL TRIAL: NCT04068948
Title: Comparing Pediatric Oral Sedation Outcomes Using Midazolam and Hydroxyzine With and Without Meperidine
Brief Title: Comparing Pediatric Dental Oral Sedation Outcomes With and Without Meperidine in Children Aged 3-7 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Travis Nelson, Clinical Associate Professor, School of Dentistry, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00006758
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Results first posted 2023-12-05 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-12

CONDITIONS: Dental Caries in Children; Pediatric Dental Sedation; Meperidine; Hydroxyzine; Midazolam
MeSH Terms: interventions — Meperidine; Hydroxyzine; Midazolam

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical trial where participants are assigned randomly to receive a sedation regimen of either midazolam+hydroxyzine+meperidine or midazolam+hydroxyzine.
Who Masked: Participant
Masking Description: The participant is unaware of the regimen given. The care provider and investigator(s) are aware of the regimen given.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Midazolam, Hydroxyzine, Meperidine (Active Comparator): Participants assigned to this group will receive a regimen of Midazolam 0.5mg/kg, Hydroxyzine 1.0mg/kg, and Meperidine 1.5mg/kg prior to their dental procedure.
  Interventions: Drug: Meperidine; Drug: Hydroxyzine; Drug: Midazolam
- Midazolam, Hydroxyzine (Experimental): Participants assigned to this group will receive a regimen of Midazolam 0.5mg/kg, and Hydroxyzine 1.0mg/kg prior to their dental procedure.
  Interventions: Drug: Hydroxyzine; Drug: Midazolam

INTERVENTIONS:
Drug: Meperidine — This intervention assesses a child's behavioral outcome for dental procedural sedation in combination with midazolam and hydroxyzine. Children participating in the study will randomly be assigned to receive either a drug regimen of midazolam+hydroxyzine, or midazolam+hydroxyzine+meperidine.
  Arms: Midazolam, Hydroxyzine, Meperidine
Drug: Hydroxyzine — This intervention is given to children for a sedative effect. Children participating in the study will randomly be assigned to receive either a drug regimen of midazolam+hydroxyzine, or midazolam+hydroxyzine+meperidine.
Drug: Midazolam — This intervention is given to children for a sedative effect. Children participating in the study will randomly be assigned to receive either a drug regimen of midazolam+hydroxyzine, or midazolam+hydroxyzine+meperidine.

SUMMARY:
The primary objective of this randomized controlled trial is to assess the effects of oral sedation using midazolam and hydroxyzine with and without meperidine (a narcotic) on sedation outcomes in pediatric dental patients undergoing dental treatment at the University of Washington Center for Pediatric Dentistry. Procedural sedation can be offered as an option for dental treatment for a young, potentially uncooperative pediatric patient to safely and effectively complete dental restorative needs. Both sedation regimens are already regularly used for patients at the UW CPD. The goal of this study is to assess if removing a narcotic from the regimen will produce the same behavioral success outcomes as a regimen with a narcotic. Our hypothesis is that patients who receive oral sedation using midazolam, hydroxyzine, and meperidine will experience fewer behavioral failures than those who receive oral sedation using midazolam and hydroxyzine without meperidine.

The secondary objective of this project is to evaluate the relationship between child temperament and sedation outcome in each treatment group.

DETAILED DESCRIPTION:
Young children in the dental setting can pose significant behavioral challenges. These patients may have dental anxiety or lack the effortful control (self-regulation) to successfully navigate the dental experience. Oral procedural sedation is an advanced pharmacological behavior guidance technique that can be used as part of the pediatric dentist's armamentarium when basic behavior guidance techniques are likely to be ineffective. Oral sedation can be a valuable tool, not only to facilitate dental treatment, but also to protect a young child's psyche, reduce dental fear, and ensure safety of both the patient and the dental team.

Case selection is crucial to optimizing sedation outcomes. In addition to biological factors like age, gender, and weight, temperament must also be carefully evaluated for the pediatric oral sedation candidate. Compared with children with high levels of effortful control, children who exhibit high levels of impulsivity may be more likely to respond poorly to uncomfortable or unfamiliar procedures, exhibit uncooperative behavior during sedation, and ultimately experience more sedation failures.

There is no standard drug regimen or protocol for oral sedation. Medications used for sedation studies often have a wide therapeutic range, and dosages used in the literature vary widely. Varying drug regimens can also be used depending on operator preference and the extent of the procedure. Benzodiazepines, opioids, and antihistamines are commonly used drug options that can be used alone or in combination to achieve desired sedative effects and minimize potential side effects of counterpart drugs. For example, midazolam is a rapid-onset, short acting benzodiazepine that offers a sedative effect with some degree of amnesia. These qualities make midazolam an ideal sedative for relatively minor or quick operative procedures in young children. An opioid such as meperidine can be added to potentiate the sedative effect and offer analgesia for lengthier, more complex procedures. Additionally, an antihistamine like hydroxyzine can be added for additional sedative effects as well as an antiemetic effect to counter potential nausea from the use of an opioid. The use of supplemental nitrous oxide/oxygen (N2O/O2) in conjunction with a chosen sedation regimen has been shown to further potentiate sedation effects and improve sedation outcomes.

Despite proving to be an effective behavior management technique, procedural sedation poses its own set of risks. Compared with intravenous or intranasal methods of drug delivery, oral delivery of sedation medications can be challenging due to longer and more variable onset to sedation, unpredictable hepatic first-pass absorption and bioavailability, and an inability to titrate the medications. Sedation effects may linger long after the procedure is completed and affect post-discharge outcomes. Additionally, the use of multiple medications has been shown to increase the risk of adverse outcomes compared with single or dual-combination drug regimens.

The majority of adverse events during sedation can be avoided with careful case selection, medication dosing, and proper intra-operative monitoring. When adverse events do occur, they are typically due to respiratory depression, and can include laryngospasm, neurologic injury, and death. Thus, to avoid oversedation and subsequent adverse sequelae, multi-drug regimens (especially those that contain opioids like meperidine) must be used judiciously.

The midazolam/meperidine/hydroxyzine regimen is a popular combination of medications for pediatric dental sedation. The increase in the use of meperidine has been associated with a movement away from utilization of chloral hydrate (another sedative with no reversal agent, previously frequently used in conjunction with a combination of the aforementioned drugs or other drugs). While there are studies comparing sedation regimens that include both chloral hydrate and meperidine used together, meperidine is an increasingly preferred option over chloral hydrate for procedural sedation, especially with the availability of a reversal agent for the opioid in the instance of oversedation, as well as a shorter half-life compared with chloral hydrate. While narcotic-containing regimens are popular, there are still inherent risks in utilization of an opioid in any sedation regimen. Several studies have been published comparing sedation regimens that include meperidine, but to date, there are no studies comparing the efficacy of midazolam and hydroxyzine with and without meperidine. Additionally, many studies compare side effects of different regimens (for example, post-operative drowsiness, nausea, time spent asleep, crying), but few utilize the Houpt Behavior Rating that we plan to use to categorize sedation outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Are between 36-95 months of age and are planned for dental treatment at the University of Washington Center for Pediatric Dentistry,
2. Are ASA I or II, (healthy, or have mild, well-controlled systemic disease)
3. Are under the 95th weight for age BMI (body mass index) percentile,
4. Are able to take diagnostic bitewing dental radiographs,
5. Are able to take medications by mouth,
6. Have Brodsky scores of II or less (tonsil sizes take up less than 50% of the oropharyngeal opening at the back of the throat),
7. Are planned to receive operative treatment under local anesthesia,
8. Can understand and communicate with providers in English.

Exclusion Criteria:

1. Are diagnosed with autism, ADHD, or any other psychiatric or behavioral diagnosis,
2. Are ASA III or higher (severe systemic disease),
3. Are above the 95th weight for age BMI percentile,
4. Are unable to take diagnostic radiographs,
5. Will not tolerate taking medications by mouth,
6. Have Brodsky scores of greater than II (tonsil sizes take up more than 50% of the oropharyngeal opening at the back of the throat),
7. Have undergone oral sedation at a previous dental appointment,
8. Cannot understand or communicate with providers in English.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Travis M Nelson, DDS, Principal Investigator — University of Washington
Locations (1):
- University of Washington Center for Pediatric Dentistry, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ashley PF, Chaudhary M, Lourenco-Matharu L. Sedation of children undergoing dental treatment. Cochrane Database Syst Rev. 2018 Dec 17;12(12):CD003877. doi: 10.1002/14651858.CD003877.pub5. PMID 30566228
- [Background] Attri JP, Sharan R, Makkar V, Gupta KK, Khetarpal R, Kataria AP. Conscious Sedation: Emerging Trends in Pediatric Dentistry. Anesth Essays Res. 2017 Apr-Jun;11(2):277-281. doi: 10.4103/0259-1162.171458. PMID 28663606
- [Background] Chicka MC, Dembo JB, Mathu-Muju KR, Nash DA, Bush HM. Adverse events during pediatric dental anesthesia and sedation: a review of closed malpractice insurance claims. Pediatr Dent. 2012 May-Jun;34(3):231-8. PMID 22795157
- [Background] Chowdhury J, Vargas KG. Comparison of chloral hydrate, meperidine, and hydroxyzine to midazolam regimens for oral sedation of pediatric dental patients. Pediatr Dent. 2005 May-Jun;27(3):191-7. PMID 16173222
- [Background] Cote CJ, Notterman DA, Karl HW, Weinberg JA, McCloskey C. Adverse sedation events in pediatrics: a critical incident analysis of contributing factors. Pediatrics. 2000 Apr;105(4 Pt 1):805-14. doi: 10.1542/peds.105.4.805. PMID 10742324
- [Background] Gentz R, Casamassimo P, Amini H, Claman D, Smiley M. Safety and Efficacy of 3 Pediatric Midazolam Moderate Sedation Regimens. Anesth Prog. 2017 Summer;64(2):66-72. doi: 10.2344/anpr-64-02-04. PMID 28604093
- [Background] Kain ZN, MacLaren J, McClain BC, Saadat H, Wang SM, Mayes LC, Anderson GM. Effects of age and emotionality on the effectiveness of midazolam administered preoperatively to children. Anesthesiology. 2007 Oct;107(4):545-52. doi: 10.1097/01.anes.0000281895.81168.c3. PMID 17893449
- [Background] Lane KJ, Nelson TM, Thikkurissy S, Scott JM. Assessing Temperament as a Predictor of Oral Sedation Success Using the Children's Behavior Questionnaire Short Form. Pediatr Dent. 2015 Sep-Oct;37(5):429-35. PMID 26531085
- [Background] McKee KC, Nazif MM, Jackson DL, Barnhart DC, Close J, Moore PA. Dose-responsive characteristics of meperidine sedation in preschool children. Pediatr Dent. 1990 Jul-Aug;12(4):222-7. PMID 2077497
- [Background] McCormack L, Chen JW, Trapp L, Job A. A comparison of sedation-related events for two multiagent oral sedation regimens in pediatric dental patients. Pediatr Dent. 2014 Jul-Aug;36(4):302-8. PMID 25197995
- [Background] Shapira J, Kupietzky A, Kadari A, Fuks AB, Holan G. Comparison of oral midazolam with and without hydroxyzine in the sedation of pediatric dental patients. Pediatr Dent. 2004 Nov-Dec;26(6):492-6. PMID 15646910

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children scheduled for dental treatment with oral moderate sedation at the University of Washington Center for Pediatric Dentistry were recruited for the study from 2019-2022
Groups:
- Midazolam, Hydroxyzine, Meperidine: Participants assigned to this group received a regimen of Midazolam 0.5mg/kg, Hydroxyzine 1.0mg/kg, and Meperidine 1.5mg/kg prior to their dental procedure.
Period: Overall Study
Arm/Group | Midazolam, Hydroxyzine, Meperidine | Midazolam, Hydroxyzine
Started | 20 | 17
Completed | 20 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Midazolam, Hydroxyzine: Participants assigned to this group received a regimen of Midazolam 0.5mg/kg, and Hydroxyzine 1.0mg/kg prior to their dental procedure.
- Total: Total of all reporting groups
Arm/Group | Midazolam, Hydroxyzine, Meperidine | Midazolam, Hydroxyzine | Total
Number analyzed (Participants) | 20 | 17 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 17 | 37
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: months] | 69.15 [38 to 93] | 69.23 [38 to 87] | 69.19 [38 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 10 | 9 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 20 | 17 | 37
Region of Enrollment [Count of Participants; unit: Participants] — Seattle, WA
  Participants
    United States | 20 | 17 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Sedation
Description: Children's behavior during sedation is rated on the Houpt Behavior Rating Scale. A successful sedation is rated as Excellent, Very Good, or Good. A failed sedation is rated as Fair, Poor, or Aborted.
Time Frame: At completion of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam, Hydroxyzine, Meperidine | Midazolam, Hydroxyzine
Number analyzed (Participants) | 20 | 17
Participants | 11 | 9

2. Secondary Outcome: Child Temperament According to CBQ-SF and Association With Sedation Outcomes
Description: Children's temperament will be assessed via parental completion of the Child Behavior Questionnaire Short Form (CBQ-SF) to assess which child temperaments may be more suitable candidates for dental oral sedation.
  The CBQ-SF is a set of 94 statements scoring a child's temperament on 15 domains: activity level, anger/frustration, approach/positive anticipation, attentional focusing, discomfort, falling reactivity/soothability, fear, high intensity pleasure, impulsivity, inhibitory control, low intensity pleasure, perceptual sensitivity, sadness, shyness, and smiling and laughter.
  There is no "better or worse outcome." The range is from 1 (minimum) to 7 (maximum) for all domains. A higher score indicates closer alignment with that temperament domain.
  Subscales of each primary domain (Effortful Control, Negative Affectivity, and Extraversion/Surgency) are combined and the sums averaged to create the total score for the 3 primary domains
Time Frame: During procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Midazolam, Hydroxyzine, Meperidine | Midazolam, Hydroxyzine
Number analyzed (Participants) | 19 | 17
score on a scale
  Effortful Control | 5.38 (0.47) | 5.84 (0.81)
  Negative Affectivity | 4.44 (0.75) | 4.12 (0.43)
  Extraversion/Surgency | 4.30 (0.46) | 4.21 (0.50)

ADVERSE EVENTS:
Time Frame: 3 years
Description: Adverse event: Any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure.
  Serious Adverse Event: Any AE that results in any of the following outcomes:
  * Death
  * Life-threatening
  * Event requiring inpatient hospitalization or prolongation of existing hospitalization
  * Persistent or significant disability/incapacity
Arm/Group | Midazolam, Hydroxyzine, Meperidine | Midazolam, Hydroxyzine
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/17
Other Adverse Events (participants affected / at risk) | 0/20 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-01-15): https://cdn.clinicaltrials.gov/large-docs/48/NCT04068948/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-15): https://cdn.clinicaltrials.gov/large-docs/48/NCT04068948/SAP_001.pdf